CLINICAL TRIAL: NCT01344538
Title: Phase II Study of the Effects of Ginger Root Extract on Eicosanoids in Colon Mucosa in People at Normal Risk for Colorectal Cancer
Brief Title: Ginger for Colorectal Cancer Prevention
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Suzanna Zick, Research Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Ginger-01HR
Record Dates: First submitted 2011-04-27; First posted 2011-04-29 (Estimated); Results first posted 2016-08-11 (Estimated); Last update posted 2016-08-11 (Estimated); Status verified 2016-06

CONDITIONS: Colorectal Cancer
Keywords: ginger; Zingiber officinale; Cancer Risk Reductive; Eicosanoids; Colorectal Cancer; Inflammation
MeSH Terms: conditions — Colorectal Neoplasms; Inflammation | interventions — ginger extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ginger Root Extract (Experimental)
  Interventions: Drug: Ginger Root Extract (Pure Encapsulations)
- Lactose Capsule (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo Capsule

INTERVENTIONS:
Drug: Ginger Root Extract (Pure Encapsulations) — 2.0 g per day (10:1 extract)
  Arms: Ginger Root Extract
Dietary Supplement: Placebo Capsule — 2.0 g per day
  Arms: Lactose Capsule

SUMMARY:
The purpose of this study is to determine if ginger root extract when taken daily for 28 days is able to decrease levels of inflammatory chemicals called eicosanoids in the gut tissue of people who are at normal risk and those at increased of developing colorectal cancer compared to people taking placebo.

ELIGIBILITY:
Inclusion Criteria Normal Risk:

* 18 years or older and in good health as defined by an unremarkable medical history, physical and screening blood work (chemistry screen, complete blood count) within 60 days of study entry.
* No chronic medication use was allowed and participants could not have taken aspirin or related NSAIDs during the study or 14 days before the first dose of the study medication.
* Participants also had to be classified as being at normal-risk for developing colorectal cancer. Normal-risk was defined as having: no first-degree relatives with colon cancer diagnosed before the age of 60; no personal history of colorectal cancer and no adenomas >1 cm in size or containing carcinoma in situ

Exclusion Criteria for both Normal and Increased Risk for Colorectal Cancer:

1. a history of peptic ulcer disease, gastrointestinal bleeding from gastric or duodenal ulcers, or gastrin secreting tumors;
2. pregnant or lactating women;
3. history of cardiovascular disease;
4. lactose intolerance;
5. or an allergy to ginger
6. a history of familial colorectal cancer syndromes;.

Inclusion Criteria Increased Risk:

* 18 years or older and in good health as defined by an unremarkable medical history, physical and screening blood work (chemistry screen, complete blood count) within 60 days of study entry.
* No chronic medication use was allowed and participants could not have taken aspirin or related NSAIDs during the study or 14 days before the first dose of the study medication.
* Participants also had to be classified as being at increased-risk for developing colorectal cancer. Increased-risk is defined as having at least one of the following: a first-degree relatives with colon cancer diagnosed before the age of 60; a personal history of early stage colorectal cancer and/or no adenomas >1 cm in size or containing carcinoma in situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-04; Primary Completion 2011-05 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanna M Zick, ND, MPH, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Zick SM, Turgeon DK, Vareed SK, Ruffin MT, Litzinger AJ, Wright BD, Alrawi S, Normolle DP, Djuric Z, Brenner DE. Phase II study of the effects of ginger root extract on eicosanoids in colon mucosa in people at normal risk for colorectal cancer. Cancer Prev Res (Phila). 2011 Nov;4(11):1929-37. doi: 10.1158/1940-6207.CAPR-11-0224. Epub 2011 Oct 11. PMID 21990307
- [Result] Citronberg J, Bostick R, Ahearn T, Turgeon DK, Ruffin MT, Djuric Z, Sen A, Brenner DE, Zick SM. Effects of ginger supplementation on cell-cycle biomarkers in the normal-appearing colonic mucosa of patients at increased risk for colorectal cancer: results from a pilot, randomized, and controlled trial. Cancer Prev Res (Phila). 2013 Apr;6(4):271-81. doi: 10.1158/1940-6207.CAPR-12-0327. Epub 2013 Jan 9. PMID 23303903
- [Result] Jiang Y, Turgeon DK, Wright BD, Sidahmed E, Ruffin MT, Brenner DE, Sen A, Zick SM. Effect of ginger root on cyclooxygenase-1 and 15-hydroxyprostaglandin dehydrogenase expression in colonic mucosa of humans at normal and increased risk for colorectal cancer. Eur J Cancer Prev. 2013 Sep;22(5):455-60. doi: 10.1097/CEJ.0b013e32835c829b. PMID 23222413
- [Derived] Zick SM, Turgeon DK, Ren J, Ruffin MT, Wright BD, Sen A, Djuric Z, Brenner DE. Pilot clinical study of the effects of ginger root extract on eicosanoids in colonic mucosa of subjects at increased risk for colorectal cancer. Mol Carcinog. 2015 Sep;54(9):908-15. doi: 10.1002/mc.22163. Epub 2014 Apr 24. PMID 24760534

RESULTS

PARTICIPANT FLOW:
Groups:
- Ginger Root Extract: Ginger Root Extract (Pure Encapsulations) : 2.0 g per day (10:1 extract)
- Lactose Capsule: Placebo Capsule : 2.0 g per day
Period: Overall Study
Arm/Group | Ginger Root Extract | Lactose Capsule
Started | 16 | 17
Completed | 14 | 16
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: 33 people enrolled with 3 withdrawn
Groups:
- Total: Total of all reporting groups
Arm/Group | Ginger Root Extract | Lactose Capsule | Total
Number analyzed (Participants) | 16 | 17 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (13.1) | 33.4 (10.1) | 34.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 7 | 9 | 16
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 33

OUTCOME MEASURES:

1. Primary Outcome: Evaluate Whether 2.0g of Ginger Taken Daily, Standardized to 5%-Gingerols for Four Weeks Will Result in Bioactive Levels in Colonic Tissue Sufficient to Reduce Mucosal Prostaglandin E2 (PGE2), a Marker of Cyclooxygenase Function Versus Placebo.
Description: % Change between baseline and day 28 in PGE2 levels standardized by protein
Time Frame: Baseline and day 28
Measure: Mean (Standard Deviation); unit: percentage of change from baseline
Arm/Group | Lactose Capsule | Ginger Root Extract
Number analyzed (Participants) | 16 | 14
percentage of change from baseline | 31.9 (89.8) | -6.7 (51.6)
Statistical Analysis 1: Comparison: Lactose Capsule vs Ginger Root Extract; Test type: Superiority or Other; p < 0.05, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Ginger Root Extract | Lactose Capsule
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/16
Other Adverse Events (participants affected / at risk) | 5/14 | 7/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ginger Root Extract (N=14) | Lactose Capsule (N=16)
Stomach upset (Gastrointestinal disorders) | 5 | 6
headache (General disorders) | 1 | 1
Fatigue (General disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No